CLINICAL TRIAL: NCT04452656
Title: Analgesic Efficacy of Ultrasound Guided Bilateral Erector Spinae Plane Block Versus Fentanyl Infusion in Pediatric Patients Undergoing Cardiac Surgeries. a Randomized Controlled Study.
Brief Title: Analgesic Efficacy of Ultrasound Guided Bilateral Erector Spinae Plane Block in Pediatric.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AHMED ALI GADO, Director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N159-2020
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia, Local; Analgesia
Keywords: Erector spinae plane block; Pediatric; sternotomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blindness will be achieved by patient codes which will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A physician not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anaesthesiologist who is expert in doing the Erector spinae plane block in patients included within the block group. This expert anaesthesiologist will not be involved in collecting data but another anaesthesia doctor will be responsible for patient management and collecting the intraoperative and postoperative data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral erector spinae plane block (Active Comparator): The patient WILL receive bilateral erector spinae plane block.
  Interventions: Procedure: bilateral erector spinae block
- NO BLOCK (No Intervention): The patient will not receive Erector spinae plane block

INTERVENTIONS:
Procedure: bilateral erector spinae block — An ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T3 spinous process corresponding to the T2 transverse process.
  Three muscles; trapezius , rhomboids major , and erector spinae will be identified superior to the hyperechoic transverse process.
  Using in-plane approach a 25 G needle will be inserted in caudal-cephalad direction, until the tip is deep to erector spinae muscle.
  Correct needle tip location will be confirmed by injecting 3 mL of saline and visualizing the linear LA spread in the fascial plane between the erector spinae muscle and the transverse process..
  0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) will be injected and visualizing the linear LA spread in the fascial plane between the erector spinae muscle andthe transverse process12.
  Arms: bilateral erector spinae plane block

SUMMARY:
This randomized, double-blinded, study aims to compare the efficacy of analgesia and any side effects of U/S guided bilateral Erector SpinaePlane block versus non-block t paediatric patients undergoing corrective cardiac surgeries.

DETAILED DESCRIPTION:
Our study will be designed to estimate and compare the analgesic effect of single shotbilatral erector spinae plane block in pediatric patients undergoing corrective cardiac surgeries versus non-block as the control group. Our primary outcome will be the total dose of intraoperative fentanyl boluses.

Randomization will be achieved by using an online random number generator. Patient codes will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A medical personnel not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anesthesiologist who is expert in doing the ESP block in patients included within the block group. The anesthesia team who managed the patients intraoperatively did not share in recording data for the research. However, another physcian will be responsible for recording the intraoperative data.

ELIGIBILITY:
Inclusion Criteria:

* Age:6 months-7 years.
* ASA, American Society of Anesthesiology, II and III .
* Patients undergoing cardiac surgeries with midline sternotomy incision.

Exclusion Criteria:

* Patients whose parents or legal guardians refusing to participate.
* Preoperative mechanical ventilation.
* Preoperative inotropic drug infusion.
* Known or suspected coagulopathy.
* Any congenital anomalies of the sacrum/the vertebral column or any infection at the site of injection.
* Known or suspected allergy to any of the studied drugs.
* Elevated liver enzymes more than the normal values.
* Renal function impairment (Creatinine value more than 1.2 mg/dl or BUN more than 20mg/dl).

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
The total dose of intraoperative fentanyl boluses in microgram. | 3 months
  The total dose of intraoperative fentanyl boluses in microgram

SECONDARY OUTCOMES:
Pain assessment at postoperatively by FLACC score | 3 months
  Pain assessment postoperatively by FLACC score
Total consumption of morphine during the first 24 hours postoperatively. | 3 monts
  Total consumption of morphine during the first 24 hours postoperatively
extubation time | 3 months
  time from finishing skin incision suturing and cessation of anesthesia to successful removal of endotracheal tube.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The patients data are confidential

REFERENCES:
- [Background] Anand VG, Kannan M, Thavamani A, Bridgit MJ. Effects of dexmedetomidine added to caudal ropivacaine in paediatric lower abdominal surgeries. Indian J Anaesth. 2011 Jul;55(4):340-6. doi: 10.4103/0019-5049.84835. PMID 22013248
- [Background] Anand KJ, Hickey PR. Halothane-morphine compared with high-dose sufentanil for anesthesia and postoperative analgesia in neonatal cardiac surgery. N Engl J Med. 1992 Jan 2;326(1):1-9. doi: 10.1056/NEJM199201023260101. PMID 1530752
- [Background] El Shamaa HA, Ibrahim M. A comparative study of the effect of caudal dexmedetomidine versus morphine added to bupivacaine in pediatric infra-umbilical surgery. Saudi J Anaesth. 2014 Apr;8(2):155-60. doi: 10.4103/1658-354X.130677. PMID 24843324
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kaushal B, Chauhan S, Magoon R, Krishna NS, Saini K, Bhoi D, Bisoi AK. Efficacy of Bilateral Erector Spinae Plane Block in Management of Acute Postoperative Surgical Pain After Pediatric Cardiac Surgeries Through a Midline Sternotomy. J Cardiothorac Vasc Anesth. 2020 Apr;34(4):981-986. doi: 10.1053/j.jvca.2019.08.009. Epub 2019 Aug 12. PMID 31515190
- [Background] Munoz F, Cubillos J, Bonilla AJ, Chin KJ. Erector spinae plane block for postoperative analgesia in pediatric oncological thoracic surgery. Can J Anaesth. 2017 Aug;64(8):880-882. doi: 10.1007/s12630-017-0894-0. Epub 2017 Apr 26. No abstract available. PMID 28447318
- [Background] De la Cuadra-Fontaine JC, Concha M, Vuletin F, Arancibia H. Continuous Erector Spinae Plane block for thoracic surgery in a pediatric patient. Paediatr Anaesth. 2018 Jan;28(1):74-75. doi: 10.1111/pan.13277. No abstract available. PMID 29226529
- [Background] Hernandez MA, Palazzi L, Lapalma J, Forero M, Chin KJ. Erector Spinae Plane Block for Surgery of the Posterior Thoracic Wall in a Pediatric Patient. Reg Anesth Pain Med. 2018 Feb;43(2):217-219. doi: 10.1097/AAP.0000000000000716. PMID 29278605
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experiences of erector spinae plane block for children. J Clin Anesth. 2018 Feb;44:41. doi: 10.1016/j.jclinane.2017.10.021. No abstract available. PMID 29100022 (Retraction: PMID 35537948 J Clin Anesth. 2022 Sep;80:110806)
- [Background] Kaplan I, Jiao Y, AuBuchon JD, Moore RP. Continuous Erector Spinae Plane Catheter for Analgesia After Infant Thoracotomy: A Case Report. A A Pract. 2018 Nov 1;11(9):250-252. doi: 10.1213/XAA.0000000000000799. PMID 29794802
- [Background] Hernandez MA, Palazzi L, Lapalma J, Cravero J. Erector spinae plane block for inguinal hernia repair in preterm infants. Paediatr Anaesth. 2018 Mar;28(3):298-299. doi: 10.1111/pan.13325. Epub 2018 Jan 17. PMID 29341379
- [Background] Merkel S, Voepel-Lewis T, Malviya S. Pain assessment in infants and young children: the FLACC scale. Am J Nurs. 2002 Oct;102(10):55-8. doi: 10.1097/00000446-200210000-00024. No abstract available. PMID 12394307